CLINICAL TRIAL: NCT00596830
Title: Randomized, Open Label, Phase III Trial Of CP- 751,871 In Combination With Paclitaxel And Carboplatin Versus Paclitaxel And Carboplatin In Patients With Non Small Cell Lung Cancer
Brief Title: Carboplatin And Paclitaxel With Or Without CP-751, 871 (An IGF-1R Inhibitor) For Advanced NSCLC Of Squamous, Large Cell And Adenosquamous Carcinoma Histology
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4021016
Record Dates: First submitted 2008-01-03; First posted 2008-01-17 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Carcinoma, Squamous Cell; Carcinoma, Adenosquamous; Carcinoma, Large Cell; Carcinoma, Non-Small-Cell Lung
Keywords: IGF-1R inhibitor; Non-small-cell lung carcinoma; CP-751; 871
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Adenosquamous; Carcinoma, Large Cell; Carcinoma, Non-Small-Cell Lung | interventions — figitumumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients in Arm A will receive CP-751, 871 in combination with paclitaxel and carboplatin intravenously every 21 days for up to six cycles.'
  Interventions: Drug: CP-751,871 (Figitumumab); Drug: Carboplatin; Drug: Paclitaxel
- B (Active Comparator): Patient in Arm B will receive paclitaxel and carboplatin intravenously every 21 days for up to six cycles.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: CP-751,871 (Figitumumab) — CP 751,871 is a potent and selective fully human monoclonal antibody against the insulin like growth factor 1 receptor (IGF-1R). Patients in Arm A will receive CP-751, 871 intravenously every 21 days for up to six cycles.
  Arms: A
Drug: Carboplatin — Carboplatin is a standard chemotherapeutic agent used in patients with lung cancer. Patients in Arm A will receive carboplatin intravenously every 21 days for up to six cycles.
  Arms: A
Drug: Paclitaxel — Paclitaxel is a standard chemotherapeutic agent used in patients with lung cancer. Patients in Arm A will receive paclitaxel intravenously every 21 days for up to six cycles.
  Arms: A
Drug: Carboplatin — Carboplatin is a standard chemotherapeutic agent used in patients with lung cancer. Patient in Arm B will receive carboplatin intravenously every 21 days for up to six cycles.
  Arms: B
Drug: Paclitaxel — Paclitaxel is a standard chemotherapeutic agent used in patients with lung cancer. Patient in Arm B will receive paclitaxel intravenously every 21 days for up to six cycles.
  Arms: B

SUMMARY:
Determine whether the addition of CP- 751,871 in combination with paclitaxel plus carboplatin prolongs survival in patients with locally advanced (Stage IIIB with pleural effusion) or metastatic (Stage IV or recurrent) NSCLC of non adenocarcinoma histology.

DETAILED DESCRIPTION:
The study was discontinued on December 29, 2009 due to an analysis by an independent Data Safety Monitoring Committee indicating that the addition of CP-751,871 [figitumumab] to paclitaxel plus carboplatin would be unlikely to meet the primary endpoint of improving overall survival compared to paclitaxel plus carboplatin alone. The DSMC recommendation to terminate the trial was based on futility, not on specific safety concerns; however, the DSMC recommended to investigate hyperglycemia as a potential contributor to the morbidity of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of non small cell lung cancer with a primary histology of predominantly squamous cell, large cell or adenosquamous carcinoma.
* Advanced NSCLC with documented Stage IIIB (with pleural effusion) or Stage IV or recurrent disease.
* No prior systemic treatment for NSCLC, except for adjuvant chemotherapy. Adjuvant chemotherapy must have completed for greater than or equal to 12 months prior to randomization.
* Prior surgery or radiation therapy is permitted if completed at least 3 weeks prior to randomization and all acute toxicities have resolved.
* ECOG performance status (PS) 0 or 1.

Exclusion Criteria:

* Patients with symptomatic central nervous system (CNS) metastases are not permitted.
* Patients requiring chronic steroid use or patients with uncontrolled diabetes are not permitted.
* Patients with other active cancer types are not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (233):
- United States (136):
  - Pfizer Investigational Site, Florence, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Muscle Shoals, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Littleton, Colorado
  - Pfizer Investigational Site, Lone Tree, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Parker, Colorado
  - Pfizer Investigational Site, Thornton, Colorado
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Norwich, Connecticut
  - Pfizer Investigational Site, Hudson, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Lake City, Florida
  - Pfizer Investigational Site, Miramar Beach, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Port Saint Lucie, Florida
  - Pfizer Investigational Site, Spring Hill, Florida
  - Pfizer Investigational Site, Alpharetta, Georgia
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Cumming, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Duluth, Georgia
  - Pfizer Investigational Site, Lake Spivey, Georgia
  - Pfizer Investigational Site, Lawrenceville, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Snellville, Georgia
  - Pfizer Investigational Site, Coeur d'Alene, Idaho
  - Pfizer Investigational Site, Arlington Heights, Illinois
  - Pfizer Investigational Site, Aurora, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Elk Grove Village, Illinois
  - Pfizer Investigational Site, Galesburg, Illinois
  - Pfizer Investigational Site, Winfield, Illinois
  - Pfizer Investigational Site, Yorkville, Illinois
  - Pfizer Investigational Site, Avon, Indiana
  - Pfizer Investigational Site, Beech Grove, Indiana
  - Pfizer Investigational Site, Hobart, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Mooresville, Indiana
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Shawnee Mission, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Lawrence, Massachusetts
  - Pfizer Investigational Site, Quincy, Massachusetts
  - Pfizer Investigational Site, Stoneham, Massachusetts
  - Pfizer Investigational Site, Weymouth, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Saint Joseph, Michigan
  - Pfizer Investigational Site, Saint Louis Park, Minnesota
  - Pfizer Investigational Site, Columbus, Mississippi
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Oxford, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lee's Summit, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Manchester, New Hampshire
  - Pfizer Investigational Site, Lake Success, New York
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, Oneida, New York
  - Pfizer Investigational Site, Oswego, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Burlington, North Carolina
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Dover, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Clairton, Pennsylvania
  - Pfizer Investigational Site, Greensburg, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, McKeesport, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Radnor, Pennsylvania
  - Pfizer Investigational Site, Sayre, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Sumter, South Carolina
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Maryville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Sam Houston, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Grapevine, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Round Rock, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, San Marcos, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Bountiful, Utah
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Provo, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Valley City, Utah
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Christiansburg, Virginia
  - Pfizer Investigational Site, Fairfax, Virginia
  - Pfizer Investigational Site, Gainesville, Virginia
  - Pfizer Investigational Site, Leesburg, Virginia
  - Pfizer Investigational Site, Roanoke, Virginia
  - Pfizer Investigational Site, Salem, Virginia
  - Pfizer Investigational Site, Winchester, Virginia
  - Pfizer Investigational Site, Woodbridge, Virginia
  - Pfizer Investigational Site, Wytheville, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Spokane Valley, Washington
- Australia (4):
  - Pfizer Investigational Site, Albury, New South Wales
  - Pfizer Investigational Site, Port Macquarie, New South Wales
  - Pfizer Investigational Site, Geelong, Victoria
  - Pfizer Investigational Site, Wodonga, Victoria
- Austria (2):
  - Pfizer Investigational Site, Linz
  - Pfizer Investigational Site, Vienna
- Brazil (3):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Higienópolis, Sao Paulo/ Brazil
  - Pfizer Investigational Site, São Paulo, São Paulo
- Bulgaria (3):
  - Pfizer Investigational Site, Sofia, Bulgaria
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Varna
- Canada (2):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Lévis, Quebec
- Czechia (4):
  - Pfizer Investigational Site, Nová Ves pod Pleší
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Pribram I
  - Pfizer Investigational Site, Pribram V
- Finland (2):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Pori
- France (8):
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Clermond-Ferrand Cedex 01
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Saint Pierre La Réunion Cedex
  - Pfizer Investigational Site, Saint-Herblain
- Germany (5):
  - Pfizer Investigational Site, Großhansdorf
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Oldenburg
- Greece (3):
  - Pfizer Investigational Site, Thessaloniki, Pylaia
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Thessaloniki
- Hong Kong (3):
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Shatin, New Territories
  - Pfizer Investigational Site, Tuenmen
- Hungary (5):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Deszk
  - Pfizer Investigational Site, Székesfehérvár
  - Pfizer Investigational Site, Szombathely
  - Pfizer Investigational Site, Törökbálint
- India (5):
  - Pfizer Investigational Site, Navrangpura / Ahmedabad, Gujarat
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, New Delhi, New Delhi
- Italy (4):
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Orbassano (TO)
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Roma
- Japan (11):
  - Pfizer Investigational Site, Kashiwa, Chiba
  - Pfizer Investigational Site, Matsuyama, Ehime
  - Pfizer Investigational Site, Gifu, Gifu
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Akashi, Hyōgo
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Osakasayama-shi, Osaka
  - Pfizer Investigational Site, Sakai-shi, Osaka
  - Pfizer Investigational Site, Chuo-Ku, Tokyo
  - Pfizer Investigational Site, Tokyo
- Poland (5):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Siedlce
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Pfizer Investigational Site, Ponce, Puerto Rico
- Russia (4):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Samara
  - Pfizer Investigational Site, Sochi
- Slovakia (3):
  - Pfizer Investigational Site, Nitra-Zobor
  - Pfizer Investigational Site, Nové Zámky
  - Pfizer Investigational Site, Poprad
- South Korea (2):
  - Pfizer Investigational Site, Gyeonggi-do
  - Pfizer Investigational Site, Seoul
- Spain (6):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Córdoba, Cordoba
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Pamplona, Navarre
  - Pfizer Investigational Site, Valencia, Valencia
- Switzerland (2):
  - Pfizer Investigational Site, Fribourg
  - Pfizer Investigational Site, Zurich
- Taiwan (3):
  - Pfizer Investigational Site, Niao Sung Hsiang, Kaohsiung Hsien
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Adana
  - Pfizer Investigational Site, Ankara
- Ukraine (5):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Sumy

REFERENCES:
- [Derived] Roeland EJ, Fintelmann FJ, Yang R, Tarasenko L, Bonomi PD. Evaluation of Weight Gain and Overall Survival of Men Versus Women With Advanced Non-Small Cell Lung Cancer. J Cachexia Sarcopenia Muscle. 2025 Dec;16(6):e70131. doi: 10.1002/jcsm.70131. PMID 41332393
- [Derived] Langer CJ, Novello S, Park K, Krzakowski M, Karp DD, Mok T, Benner RJ, Scranton JR, Olszanski AJ, Jassem J. Randomized, phase III trial of first-line figitumumab in combination with paclitaxel and carboplatin versus paclitaxel and carboplatin alone in patients with advanced non-small-cell lung cancer. J Clin Oncol. 2014 Jul 1;32(19):2059-66. doi: 10.1200/JCO.2013.54.4932. Epub 2014 Jun 2. PMID 24888810
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021016&StudyName=Carboplatin%20And%20Paclitaxel%20With%20Or%20Without%20CP-751%2C%20871%20%28An%20IGF-1R%20Inhibitor%29%20%20For%20Advanced%20NSCLC%20Of%20Squamous%2C%20Large%20Cell%20And%20A

RESULTS

PARTICIPANT FLOW:
Groups:
- Figitumumab + Paclitaxel and Carboplatin: Figitumumab (figi, [CP-751, 871]) was given in combination with paclitaxel (200 milligram/square metre [mg/m^2]) and carboplatin (area under the concentration-time curve [AUC]=6) administered in 3-week cycles. Figi 20 milligram/kilogram (mg/kg) was administered intravenously (IV) on Day 1 of a 3-week cycle for up to 6 cycles, followed by single agent figi maintenance in every 3-week cycles after completion or discontinuation of chemotherapy for reasons other than disease progression.
- Paclitaxel and Carboplatin (Chemo): Standard platinum-based doublet chemotherapy (chemo) consisting of paclitaxel (200 milligram/square metre [mg/m^2]) and carboplatin (area under the concentration-time curve [AUC]=6) was administered via IV on Day 1 of a 3-week cycle. Chemo treatment continued for a maximum of 6 cycles.
Period: Overall Study
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Started | 342 (1 participant in this group only received paclitaxel and carboplatin (chemo).) | 339
Treated | 339 (1 participant in this group only received chemo and did not complete due to death.) | 332
Completed | 0 | 0
Not Completed | 342 | 339
Not completed — Death | 258 | 247
Not completed — Lost to Follow-up | 7 | 11
Not completed — Withdrawal by Subject | 22 | 12
Not completed — Study terminated by sponsor | 51 | 62
Not completed — Follow-up was discontinued | 1 | 0
Not completed — Randomized but not treated | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo) | Total
Number analyzed (Participants) | 342 | 339 | 681
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.0) | 61.8 (9.1) | 61.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 79 | 160
  Male | 261 | 260 | 521

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was the duration from randomization to death. For participants who are alive, overall survival was censored at the last contact.
Time Frame: Baseline until death, assessed monthly after end of treatment, up to 30 months
Population: All randomized participants where participants were classified according to the randomized treatment regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 342 | 339
months | 8.6 [7.4 to 9.3] | 9.8 [8.6 to 10.9]
Statistical Analysis 1: Comparison: Figitumumab + Paclitaxel and Carboplatin vs Paclitaxel and Carboplatin (Chemo); Test type: Superiority or Other; p = 0.064, Log Rank — The p-value stated is the 2-sided p-value from the log rank test stratified by gender, prior adjuvant chemotherapy, and histology; Hazard Ratio (HR) = 1.179, 95% CI 2-sided [0.990 to 1.404]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to first progression or death due to any cause, whichever came first. Participants last known to be alive and progression-free, with baseline and >=1 on-study assessment, were censored at last disease assessment verifying lack of progression. Progression was determined by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 (20% increase in the sum of target lesions' longest diameter over nadir, unequivocal progression of non-target disease, or appearance of new lesions).
Time Frame: At baseline, every 6 weeks until radiological disease progression or the participant begins a subsequent anticancer therapy, up to 22.7 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 342 | 339
months | 4.7 [4.2 to 5.4] | 4.6 [4.2 to 5.4]
Statistical Analysis 1: Comparison: Figitumumab + Paclitaxel and Carboplatin vs Paclitaxel and Carboplatin (Chemo); Test type: Superiority or Other; p = 0.270, Log Rank — 2-sided p-value is from the unstratified log-rank test; Hazard Ratio (HR) = 1.103, 95% CI 2-sided [0.925 to 1.315] — HR was based on the Cox proportional hazards model

3. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based on assessment of confirmed complete response (CR) or confirmed partial response(PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR defined as complete disappearance of all target lesions and non-target disease. No new lesons. PR defined as ≥30% decrease under baseline of the sum of diameters of all target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: At baseline, every 6 weeks until radiological disease progression has been documented or the participant begins a subsequent anticancer therapy, up to 22.7 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 342 | 339
percentage of participants | 33.0 [28.1 to 38.3] | 34.5 [29.5 to 39.8]
Statistical Analysis 1: Comparison: Figitumumab + Paclitaxel and Carboplatin vs Paclitaxel and Carboplatin (Chemo); Test type: Superiority or Other; p = 0.685, Chi-squared; Risk difference = -1.472, 95% CI 2-sided [-8.6 to 5.6] — Risk difference confidence interval was calculated based on a normal distribution

4. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Day 1 of every cycle (3-week cycle), every 3 weeks during maintenance phase and at the End of Treatment Visit, assessed up to 37.4 months
Population: Due to futility, the study was terminated early; therefore these data were not analyzed.
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC), Quality of Life Questionnaire-Lung Cancer 13 (QLQ- LC13) Score
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, and medicine for pain). Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: as for outcome 4
Population: Due to futility, the study was terminated early; therefore these data were not analyzed.
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range of -0.594 to 1; higher score indicates a better health state.
Time Frame: Day 1 of every cycle (3-weeks cycle), every 3 weeks during maintenance phase and at the End of Treatment Visit, assessed up to 37.4 months
Population: Due to futility, the study was terminated early; therefore EQ-5D data were not analyzed.
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Figitumumab
Time Frame: Cycle 1, Day 1 (predose and 1 hour after end of infusion); Day 1 of Cycles 2, 4, 6 (predose); Cycle 5 Day 1 (predose, 1 hour after end of infusion); 28 days and 150 days after the last figi dose
Population: This study was terminated early due to futility. As such, Cmax was not summarized.
Arm/Group | Figitumumab + Paclitaxel and Carboplatin
Number analyzed (Participants) | 0

8. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin)for Figitumumab
Time Frame: as for outcome 7
Population: This study was terminated early due to futility. As such, Cmin was not summarized.
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Total Anti-drug Antibodies (ADA)
Description: ADAs are immunogenicity indicators to figitumumab. Participants reporting positive for ADAs are indicated by an endpoint titer of no less than 6.64.
Time Frame: Cycles 1, 2, and 4 (predose); 28 days and 150 days after the last figi dose
Population: All participants who received figitumumab (CP-751,871).
Measure: Number; unit: participants
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 332 | 32
participants | 2 | 0

10. Secondary Outcome: Change From Baseline in Serum Insulin Growth Factor 1 (IGF1) Levels
Time Frame: Cycles 1 and 4 (predose) and at end of treatment
Population: This study was terminated early due to futility. As such, these data were not analyzed.
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Distinct events are presented. An event may be categorized as serious in 1 subject and as nonserious in another, or 1 subject may have experienced both kinds of events. The 1 participant who was randomized to receive figi and chemo but was treated only with chemo is included under the chemo group. Only treated participants are included.
Arm/Group | Figitumumab + Paclitaxel and Carboplatin | Paclitaxel and Carboplatin (Chemo)
Serious Adverse Events (participants affected / at risk) | 223/338 | 170/333
Other Adverse Events (participants affected / at risk) | 316/338 | 303/333
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab + Paclitaxel and Carboplatin (N=338) | Paclitaxel and Carboplatin (Chemo) (N=333)
Anaemia (Blood and lymphatic system disorders) | 2 | 9
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 11
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5
Angina pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 3 | 1
Cardiotoxicity (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Glossitis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 11 | 2
Chest pain (General disorders) | 3 | 0
Condition aggravated (General disorders) | 1 | 0
Death (General disorders) | 3 | 3
Disease progression (General disorders) | 115 | 90
Drug intolerance (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 8 | 5
Malaise (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 1 | 0
Pain (General disorders) | 3 | 3
Performance status decreased (General disorders) | 1 | 2
Pyrexia (General disorders) | 4 | 4
Sudden death (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bone abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 21 | 12
Pseudomonas infection (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 4 | 0
Septic shock (Infections and infestations) | 3 | 1
Sputum purulent (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose increased (Investigations) | 1 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 15 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Genitourinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Convulsion (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Neurotoxicity (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 0
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Arteritis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Haemorrhage (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 3 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab + Paclitaxel and Carboplatin (N=338) | Paclitaxel and Carboplatin (Chemo) (N=333)
Anaemia (Blood and lymphatic system disorders) | 93 | 85
Leukopenia (Blood and lymphatic system disorders) | 18 | 33
Neutropenia (Blood and lymphatic system disorders) | 74 | 78
Thrombocytopenia (Blood and lymphatic system disorders) | 60 | 49
Constipation (Gastrointestinal disorders) | 60 | 61
Diarrhoea (Gastrointestinal disorders) | 95 | 45
Dysphagia (Gastrointestinal disorders) | 18 | 9
Nausea (Gastrointestinal disorders) | 132 | 101
Stomatitis (Gastrointestinal disorders) | 30 | 10
Vomiting (Gastrointestinal disorders) | 82 | 46
Asthenia (General disorders) | 71 | 59
Chest pain (General disorders) | 45 | 34
Fatigue (General disorders) | 112 | 85
Mucosal inflammation (General disorders) | 27 | 9
Oedema peripheral (General disorders) | 10 | 24
Pyrexia (General disorders) | 26 | 33
Weight decreased (Investigations) | 65 | 29
Decreased appetite (Metabolism and nutrition disorders) | 128 | 75
Dehydration (Metabolism and nutrition disorders) | 28 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 74 | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 17 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 57
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 44
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 23
Dizziness (Nervous system disorders) | 37 | 32
Dysgeusia (Nervous system disorders) | 26 | 13
Headache (Nervous system disorders) | 37 | 22
Neuropathy peripheral (Nervous system disorders) | 63 | 56
Paraesthesia (Nervous system disorders) | 29 | 35
Peripheral sensory neuropathy (Nervous system disorders) | 40 | 50
Anxiety (Psychiatric disorders) | 17 | 17
Insomnia (Psychiatric disorders) | 32 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 59
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 | 65
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 32 | 21
Alopecia (Skin and subcutaneous tissue disorders) | 138 | 146
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 18
Rash (Skin and subcutaneous tissue disorders) | 28 | 20

LIMITATIONS AND CAVEATS:
The study was terminated early due to futility. CP-751,871 will not undergo further development in the indication of advanced non-adenocarcinoma non-small cell lung cancer (NSCLC).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.